CLINICAL TRIAL: NCT02436109
Title: Ultrasound Guidance for Epidural Analgesia and Anesthesia
Status: Terminated | Type: Observational
Why Stopped: study device broke
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H14-01152
Record Dates: First submitted 2015-03-31; First posted 2015-05-06 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Epidural Space Depth
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study group: elective cesarean delivery patients
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Parturients backs will be scanned using 3D ultrasound to measure the depth to the epidural space

SUMMARY:
Most women delivering by cesarean at BC Women's receive regional anesthesia; which includes spinal, epidural, or combined spinal-epidural anesthesia. In all these techniques a needle is placed in the lower back and local anesthetic is injected to freeze the body. Normally, before the needle is placed in a patients' back, the anesthesiologist will feel between their back bones with his/her fingers to find the right spot for the needle. This study will be evaluating if the distance from the skin to the appropriate spinal space measured with a novel 3D Ultrasound will equal the actual depth of the needle insertion.

DETAILED DESCRIPTION:
The investigators will be evaluating if the distance from the skin to the appropriate spinal space measured with a novel 3D Ultrasound will equal the actual depth of the needle insertion.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancy
* elective cesarean

Exclusion Criteria:

* scoliosis
* high bmi

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
epidural space depth | intraoperative
  comparison of ultrasound measured epidural space to actual needle insertion

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada